CLINICAL TRIAL: NCT02929589
Title: Ibuprofen to Decrease Opioid Use and Post-operative Pain Following Unilateral Inguinal Herniorrhaphy: A Prospective, Placebo-Controlled, Double-Blind, Randomized Controlled Trial
Brief Title: Ibuprofen to Decrease Opioid Use and Post-operative Pain Following Unilateral Inguinal Herniorrhaphy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The use of robotic surgery made this study obsolete.
Sponsor: Mike O'Callaghan Military Hospital (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FWH20160095H
Record Dates: First submitted 2016-10-04; First posted 2016-10-11 (Estimated); Results first posted 2024-03-26 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Pain; Hernia
MeSH Terms: conditions — Pain; Hernia | interventions — Ibuprofen; Opiate Substitution Treatment

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Opioid naïve patients-Group A (Experimental): Group A: Subjects will be prescribed ibuprofen 800 milligrams by mouth every 8 hours as needed for pain for 5 days, and 1 to 2 tablets of oxycodone/acetaminophen 5 milligrams/325 milligrams (Qty. 30) by mouth every 4 hours as needed for pain for 5 days.
  .
  Interventions: Drug: Ibuprofen
- Non-Opioid naïve patients-Group C (Experimental): Group C: Subjects will be prescribed ibuprofen 800 milligrams by mouth every 8 hours as needed for pain for 5 days, in addition to their preferred opioid medication prescription.
  Interventions: Drug: Ibuprofen + Opioid medication
- Opioid naïve patients-Group B (Placebo Comparator): Group B:Subjects will be prescribed 800 milligrams of a placebo pill (containing corn starch) to be taken by mouth every 8 hours as needed for pain and 1 to 2 tablets of oxycodone/acetaminophen 5 milligrams/325 milligrams (Qty. 30) by mouth every 4 hours as needed for pain for 5 days.
  Interventions: Drug: Placebo
- Non-Opioid naïve patients-Group D (Experimental): Group D: Subjects will be prescribed or advised to continue to take only their preferred current oral opioid prescription (codeine, hydrocodone, hydromorphone, morphine, methadone, oxymorphone, or transdermal fentanyl).
  Interventions: Drug: Opioid Medication

INTERVENTIONS:
Drug: Ibuprofen — ibuprofen 800 milligrams by mouth every 8 hours as needed for pain for 5 days
  Arms: Opioid naïve patients-Group A
Drug: Opioid Medication — 1 to 2 tablets of oxycodone/acetaminophen 5 milligrams/325 milligrams (Qty. 30) by mouth every 4 hours as needed for pain for 5 days
  Arms: Non-Opioid naïve patients-Group D
Drug: Placebo — 800 milligrams of a placebo pill (containing corn starch) to be taken by mouth every 8 hours as needed for pain
  Arms: Opioid naïve patients-Group B
Drug: Ibuprofen + Opioid medication — ibuprofen 800 milligrams by mouth every 8 hours as needed for pain for 5 days. 1 to 2 tablets of oxycodone/acetaminophen 5 milligrams/325 milligrams (Qty. 30) by mouth every 4 hours as needed for pain for 5 days
  Arms: Non-Opioid naïve patients-Group C

SUMMARY:
This is a prospective, randomized, double-blinded, and placebo-controlled trial comparing oxycodone/acetaminophen prescribed with or without ibuprofen for pain control following open unilateral inguinal hernia repair, with allowed exception of any currently prescribed opioid (codeine, hydrocodone, hydromorphone, morphine, methadone, oxymorphone, transdermal fentanyl), which can be continued. The patients will not be allowed to continue any over-the-counter pain medications, such as ibuprofen, naproxen, or acetaminophen containing medications, that were not prescribed by the investigators during this study. Patients not receiving Ibuprofen will be given a placebo pill composed of corn starch. The placebo pill will be formulated into the same shape, size and color as the ibuprofen capsule. Neither the investigators nor the research subjects will know if the subject is receiving a placebo versus Ibuprofen. The subjects will complete pain level and medication diaries, and will be followed for 2 months after their surgery. The research aims to discover the appropriate amount of opioid medication to prescribe to patients undergoing an elective open inguinal hernia repair, and reduce the total opioid dose needed by utilizing ibuprofen in combination. The investigators expect that the subjects who take ibuprofen will use less oxycodone/acetaminophen, and have comparable or lower mean pain levels. This could contribute to reducing the surplus opioids prescribed by physicians after surgery, which can lead to opioid use disorders. This particular procedure is common in men, and the findings have the potential to decrease the symptoms and pain of Active Duty members and DoD beneficiaries who undergo an inguinal hernia repair, and are at risk for prescription drug abuse or dependence.

DETAILED DESCRIPTION:
Screening Visit:

Discuss the purpose of the study and the required completion of study-related questionnaires and their potential impact for active duty members. (research-driven) Obtain signed Informed Consent Document and HIPAA Authorization (research-driven).

Review the patient's past medical history in Armed Forces Health Longitudinal Technology Application (AHLTA) or ESSENTRIS to verify the inclusion/exclusion criteria. (research-driven) The investigators will record the subject's tobacco use history, alcohol use history, marijuana use history, other illicit drug use history, and previous non-prescription use of opioids. (standard of care) Obtain an overall pain score, from 0 to 100, with 100 being the worst pain imaginable. (research-driven) Obtain a localized pain score from 0 to 100, with 100 being the worst pain imaginable, which the patient attributes specifically to the hernia that is scheduled for surgical intervention. (research-driven) Instruct patients to discontinue use of any over-the-counter pain medications, such as ibuprofen, naproxen, or acetaminophen containing medications, that were not prescribed by the investigators during this study.

Subjects will have the following blood test drawn, which include (research-driven):

Fasting comprehensive metabolic panel (liver function, renal function, plasma glucose tests) via 1 venipuncture (5-10 milliliters, approximately 1-2 teaspoons of blood will be drawn) Subject's CMP results must be within 30 days of the day of surgery or it will need to be repeated.

Women of childbearing potential will have a serum pregnancy test (5-10 milliliters, approximately 1-2 teaspoons of blood) or urine pregnancy test (10 drops or less than 1 milliliter of urine) (research-driven). Visit 1 (may occur the same day as the screening visit or the same day as visit 2):

The standard of care local anesthesia used for this type of surgery is bupivacaine. The surgeon will be reminded via a note in the medical record. (standard of care) Subjects will be randomized by the MOFMC Pharmacy into one of two naturally stratified groups (e.g., opioid naive patients and non-opioid naive patients), with further randomization into an opioid + ibuprofen study group or an opioid + placebo study group The MOFMC Pharmacy staff will maintain a key that can be used to un-blind the randomization scheme if needed for an emergent patient care issue. Study ID numbers will be used to maintain blinding and confidentiality. (research-driven)

Opioid naive patients (used an opioid for less than 14 days in the past 6 months, and no history of opioid use disorder at any time) will be randomized into one of two groups:

Group A: Subjects will be prescribed ibuprofen 800 milligrams by mouth every 8 hours as needed for pain for 5 days, and 1 to 2 tablets of oxycodone/acetaminophen 5 milligrams/325 milligrams (Qty. 30) by mouth every 4 hours as needed for pain for 5 days.

Group B: Subjects will be prescribed 800 milligrams of a placebo pill (containing corn starch) to be taken by mouth every 8 hours as needed for pain and 1 to 2 tablets of oxycodone/acetaminophen 5 milligrams 325 milligrams (Qty. 30) by mouth every 4 hours as needed for pain for 5 days.

Non-Opioid naive patients (opioid use for more than 14 days in the past 6 months, or history of opioid use disorder) will be randomized into one of two groups:

Group C: Subjects will be prescribed ibuprofen 800 milligrams by mouth every 8 hours as needed for pain for 5 days, in addition to their preferred opioid medication prescription.

Group D: Subjects will be prescribed or advised to continue to take only their preferred current oral opioid prescription (codeine, hydrocodone, hydromorphone, morphine, methadone, oxymorphone, or transdermal fentanyl).

Subjects will complete the Beck Depression Inventory-II or the Patient Health Questionnaire (PHQ-9) depression screen, and it will be reviewed on the same day of completion. (research-driven) Subjects will complete the Pre-Operative Activities Assessment Scale (AAS), and it will be reviewed on the same day of completion. (research-driven) Subjects will complete the Opioid Risk Tool (ORT) , and it will be reviewed on the same day of completion. (research-driven) Subjects will be asked "How likely do you think it is that you will develop an addiction problem from pain medication you take after surgery?" and chose from 1 of 4 answers: 1: "not at all"; 2: "unlikely"; 3: "somewhat likely"; or 4: "very likely". (research-driven) Subjects will be asked "On a scale of 0-100, with 0 being no pain and 100 being the worst pain imaginable, what is your average level of pain at rest in the past 24 hours?" (research-driven) Subjects will be asked "On a scale of 0-100, with 0 being no pain and 100 being the worst pain imaginable, what was your lowest level of pain when at rest in the past 24 hours? (research-driven) Subjects will be asked "On a scale of 0-100, with 0 being no pain and 100 being the worst pain imaginable, what was your highest level of pain when at rest in the past 24 hours? (research-driven) Subjects will be given a Medication and Pain Level Diary and will be instructed to complete it every day for 14 days beginning after their surgery. The investigators will record information from the subjects' surgery, for example: the start and end times of surgery and anesthesia, how long the surgery lasted, how difficult the surgery was, were the ilioinguinal, genitofemoral, or iliohypogastric nerves identified and were they protected, injured, or transected, and which opioids the anesthesiologist gives at any point during the case after incision. (research-driven) The preoperative instructions will include standardized verbal and written instructions: "After your surgery, it is expected that the patient will experience a certain amount of pain for a short period of time. The patient will be prescribed pain medication that you should take only when you are in pain. If the patient is no longer experiencing pain, the patient should stop taking the medication. If the patient does not require all of the pain medication that was prescribed, the patient should record the amount of medication that was unused and then properly dispose of the remainder." (standard of care)

Visit 2 (day of surgery-prior to surgery):

Subjects will receive prescriptions for medications according to their randomization group. These prescriptions will be filled at the MOFMC pharmacy, which will perform the subjects' randomization assignments. The ibuprofen and placebo capsules will be delivered to the MOFMC Pharmacy after being compounded by Solutions Specialty Pharmacy. (research-driven) Subjects will complete the Pre-Operative AAS (approximately 5 minutes to complete), and it will be reviewed on the same day of completion. (research-driven) Research staff will record the start and end times of the surgery, record the amounts of standard of care pain medications used during their hospital stay, document any standard of care pain assessments that were performed, and document the anesthesia the subject received. (research-driven) Subjects will be reminded in the Post Anesthesia Care Unit (PACU) to complete their Medication and Pain Level Diary and reminded to complete it every day for the 60 days beginning after they are discharged from the hospital. (research-driven)

Visit 3 (Post-Op day 0 Contact (at time of discharge from post-anesthesia care unit)):

Subjects will be contacted by research team in person or via telephone and asked the following questions in this order (research-driven):

On a scale of 0-100, with 0 being no pain and 100 being the worst pain imaginable, what is the average level of pain when at rest in the past 24 hours? On a scale of 0-100, with 0 being no pain and 100 being the worst pain imaginable, what was the lowest level of pain when at rest in the past 24 hours? On a scale of 0-100, with 0 being no pain and 100 being the worst pain imaginable, what was the highest level of pain when at rest in the past 24 hours? What pain medications are the patient taking including the strength (in milligrams), and how many total doses have you taken since your surgery? Time of last opioid medication taken? Relief from starting pain is: 0 = none, 1= a little, 2 = some, 3 = a lot, 4 = complete Subjects will be reminded to complete their Medication and Pain Level Diary. (research-driven)

Visits 4-8 (Post-op Day 1 through Day 5 Contact (each visit every 24 hours plus or minus 4 hours visit window):

Subjects will be contacted by research team in person or via telephone and asked the following questions in this order (research-driven):

On a scale of 0-100, with 0 being no pain and 100 being the worst pain imaginable, what is the average level of pain when at rest in the past 24 hours? On a scale of 0-100, with 0 being no pain and 100 being the worst pain imaginable, what was the lowest level of pain when at rest in the past 24 hours? On a scale of 0-100, with 0 being no pain and 100 being the worst pain imaginable, what was the highest level of pain since when at rest in the past 24 hours? What pain medications have been taken, including the strength (in milligrams), and how many total doses have been taken since the last study visit? Time of last opioid medication taken? Relief from starting pain is: 0 = none, 1= a little, 2 = some, 3 = a lot, 4 = complete Subjects will complete the Post-Operative AAS, and it will be reviewed on the same day of completion. (research-driven) Subjects will be reminded to complete their Medication and Pain Level Diary. (research-driven)

Visit 9 (Post-Op day 14 Contact (plus or minus 2 day visit window)):

Subjects will be contacted by research team in person or via telephone at their Post-Operative Follow Up Visit and asked the following questions in this order (in-person) (research-driven):

On a scale of 0-100, with 0 being no pain and 100 being the worst pain imaginable, what is the average level of pain when at rest in the past 24 hours? On a scale of 0-100, with 0 being no pain and 100 being the worst pain imaginable, what was your lowest level of pain since your when at rest in the past 24 hours? On a scale of 0-100, with 0 being no pain and 100 being the worst pain imaginable, what was your highest level of pain since your when at rest in the past 24 hours? What pain medications are being taken including the strength (in milligrams), and how many total doses have been taken since the last study visit? Time of last opioid medication taken? Relief from starting pain is: 0 = none, 1= a little, 2 = some, 3 = a lot, 4 = complete Subjects will complete the Post-Operative AAS, and it will be reviewed on the same day of completion. (research-driven).

Subjects will return their Medication and Pain Level Diary and be issued a new one for the remainder of the study. (research-driven) Subjects will be reminded of the two remaining contacts. (research-driven)

Visit 10 (Post-Op day 30 Contact (plus or minus 5 day visit window)):

Subjects will be contacted by research team in person or via telephone and asked the following questions in this order (research-driven):

On a scale of 0-100, with 0 being no pain and 100 being the worst pain imaginable, what is the average level of pain when at rest in the past 24 hours? On a scale of 0-100, with 0 being no pain and 100 being the worst pain imaginable, what was the lowest level of pain when at rest in the past 24 hours? On a scale of 0-100, with 0 being no pain and 100 being the worst pain imaginable, what was the highest level of pain when at rest in the past 24 hours? What pain medications are being taken including the strength (in milligrams), and how many total doses have been taken since your last study visit? Time of last opioid medication taken? Relief from starting pain is: 0 = none, 1= a little, 2 = some, 3 = a lot, 4 = complete Subjects will complete the Post-Operative AAS, and it will be reviewed on the same day of completion. (research-driven).

Subjects will be reminded to complete their Medication and Pain Level Diary. (research-driven)

Visit 11 (Post-Op day 60 Contact (plus or minus 5 day visit window)):

Subjects will be contacted by research team in person or via telephone and asked the following questions in this order (research-driven):

On a scale of 0-100, with 0 being no pain and 100 being the worst pain imaginable, what is your average level of pain when at rest in the past 24 hours? On a scale of 0-100, with 0 being no pain and 100 being the worst pain imaginable, what was the lowest level of pain since your when at rest in the past 24 hours? On a scale of 0-100, with 0 being no pain and 100 being the worst pain imaginable, what was the highest level of pain when at rest in the past 24 hours? What pain medications are being taken including the strength (in milligrams), and how many total doses have been taken since the last study visit? Time of last opioid medication taken? Relief from starting pain is: 0 = none, 1= a little, 2 = some, 3 = a lot, 4 = complete Was there a diagnosis of post-operative neuralgia at any point following your surgery? Was there a diagnosis of an inguinal hernia recurrence at any point following your surgery? Was there a diagnosis of a surgical site infection at any point following your surgery? Subjects will complete the Post-Operative AAS, and it will be reviewed on the same day of completion. (research-driven).

The Medication and Pain Level Diary will not be collected from the patient. (research-driven)

ELIGIBILITY:
PATIENTS MUST HAVE MILITARY INSURANCE TO PARTICIPATE

Inclusion/exclusion criteria:

Inclusion:

* Active Duty members and DoD beneficiary patient 18 years or older
* Elective, open unilateral inguinal herniorrhaphy using Lichtenstein (tension free with mesh) hernia repair technique Agree to take only the prescribed oral analgesic medication (oxycodone/acetaminophen), plus or minus ibuprofen, for the initial fourteen-day post-operative period, with allowed exception of any currently prescribed opioid (codeine, hydrocodone, hydromorphone, morphine, methadone, oxymorphone, transdermal fentanyl), which can be continued.Agree to honestly complete a depression screening questionnaire, illicit drug use personal history and questionnaire, and physical activity assessment questionnaire, with the knowledge that if the patient is an active duty member, this information could result in a referral to medical or command authorities for potential Uniform Code of Military Justice (UCMJ) violations or concerns for subject health and fitness for duty.

Exclusion:

* Subjects who are pregnant or nursing.
* Patients who refuse to complete the illicit drug use, physical activity, and depression questionnaires.
* Strangulated, incarcerated, or otherwise emergent, urgent, and non-elective inguinal herniorrhaphy.
* Those patients who are allergic to, refuse to take, or are otherwise unable to take oxycodone, ibuprofen, or acetaminophen medication orally for post-operative pain management.
* Patients on pain contracts, or under the care of a pain medicine specialist for management of chronic pain at the time of surgery.
* Subjects with serum creatinine level > 1.3 mg/dL as measured at the baseline study visit.
* Subjects with serum aspartate transaminase (AST) greater than 3 times the upper limit of normal (level >102 U/L)
* Subjects with serum alanine transaminase (ALT) greater than 3 times the upper limit of normal (level > 165 U/L)
* Subjects who do not speak, read, and write fluently in English.
* Subjects with a history of cirrhosis.
* Subjects enrolled in another clinical trial during the same period as their involvement as this study.
* Subjects, who in the investigator's opinion, will be unable to complete a pain diary or follow-up visits, or otherwise not comply with the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-07-05 (Actual); Primary Completion 2021-08-23 (Actual); Study Completion 2021-08-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Mike O'Callaghan Federal Medical Center, Nellis Air Force Base, Nevada, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment stopped at 18/160 as advent of robotic arm surgery made this study obsolete.
Groups:
- Opioid naïve Patients-Group A: Group A: Subjects will be prescribed ibuprofen 800 milligrams by mouth every 8 hours as needed for pain for 5 days, and 1 to 2 tablets of oxycodone/acetaminophen 5 milligrams/325 milligrams (Qty. 30) by mouth every 4 hours as needed for pain for 5 days.
  .
  Ibuprofen: ibuprofen 800 milligrams by mouth every 8 hours as needed for pain for 5 days
Period: Overall Study
Arm/Group | Opioid naïve Patients-Group A | Non-Opioid naïve Patients-Group C | Opioid naïve Patients-Group B | Non-Opioid naïve Patients-Group D
Started | 11 | 0 | 7 | 0
Completed | 8 | 0 | 7 | 0
Not Completed | 3 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Not completed — Physician Decision | 2 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Study was terminated before any subject data collected could be analyzed. Raw data are reported. No data collected was analyzed by a biostatistician.
Groups:
- Total: Total of all reporting groups
Arm/Group | Opioid naïve Patients-Group A | Non-Opioid naïve Patients-Group C | Opioid naïve Patients-Group B | Non-Opioid naïve Patients-Group D | Total
Number analyzed (Participants) | 11 | 0 | 7 | 0 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 0 | 5 | 0 | 13
  >=65 years | 3 | 0 | 2 | 0 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 2 | 0 | 2
  Male | 11 | 0 | 5 | 0 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 2 | 0 | 2
  White | 11 | 0 | 5 | 0 | 16
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Total Milligram Morphine Equivalent (MME) Units
Description: The primary outcome measure was milligram morphine equivalent units to measure pain intensity difference and total pain relief.
Time Frame: 60 days post-operation
Population: No populations were analyzed as study was terminated as obsolete after the development and use of robotic arms during surgery. Any data collected was not analyzed by a biostatistician. Raw data are reported for 15 subjects. 3/15 were screenfails in Group A.
Measure: Mean (Full Range); unit: milligram morphine equivalence units
Arm/Group | Opioid naïve Patients-Group A | Non-Opioid naïve Patients-Group C | Opioid naïve Patients-Group B | Non-Opioid naïve Patients-Group D
Number analyzed (Participants) | 8 | 0 | 7 | 0
milligram morphine equivalence units | 72 [0 to 207] |  | 88 [0 to 340] |

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for the duration of the study (screening to 60 days post-operation). Adverse events were collected as long as the subject was enrolled in the study; this depended on when surgeries were scheduled and performed.
Arm/Group | Opioid naïve Patients-Group A | Non-Opioid naïve Patients-Group C | Opioid naïve Patients-Group B | Non-Opioid naïve Patients-Group D
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/0 | 0/7 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/0 | 0/7 | 0/0
Other Adverse Events (participants affected / at risk) | 1/11 | 0/0 | 0/7 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Opioid naïve Patients-Group A (N=11) | Non-Opioid naïve Patients-Group C (N=0) | Opioid naïve Patients-Group B (N=7) | Non-Opioid naïve Patients-Group D (N=0)
Adverse Event (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Subject had stomach cramps and decrease in bowel movements. He increased dietary fiber and took prescribed Colace and it resolved. Unclear if cause was surgery or study medications. These risks are in the Protocol and ICD as likely and not serious.

LIMITATIONS AND CAVEATS:
This study was terminated early as the advent of the use of robotic surgery made this study obsolete.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-07-27): https://cdn.clinicaltrials.gov/large-docs/89/NCT02929589/Prot_SAP_001.pdf
  • Informed Consent Form (2020-07-27): https://cdn.clinicaltrials.gov/large-docs/89/NCT02929589/ICF_000.pdf